CLINICAL TRIAL: NCT03525873
Title: A Study of Cancer Related Fatigue in Patients With Metastatic Cancer Receiving Anti-PD1 Immunotherapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2017-0913; NCI-2018-00698 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0913 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-05-02; First posted 2018-05-16 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Advanced Malignant Neoplasm; Metastatic Malignant Neoplasm; Recurrent Malignant Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence | interventions — Methylphenidate; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARM I (methylphenidate, physical activity) (Experimental): Patients receive methylphenidate PO BID for up to 2 weeks in the absence of disease progression or unacceptable toxicity. Patients also complete physical activity consisting of walking and resistance exercise over 25-40 minutes QD 4 days a week. After 2 weeks, patients may continue methylphenidate at the discretion of the treating physician for up to 12 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Methylphenidate; Other: Physical Activity; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- ARM II (placebo, physical activity) (Placebo Comparator): Patients receive a matched placebo PO BID and complete physical activity as in Arm I. Treatment continues for up to 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Physical Activity; Other: Placebo; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Methylphenidate — Given PO
  Other Names: Daytrana
  Arms: ARM I (methylphenidate, physical activity)
Other: Physical Activity — Participate in physical activity
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: ARM II (placebo, physical activity)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial studies how well methylphenidate and physical activity works in reducing cancer-related fatigue in patients who are receiving anti-PD1 immunotherapy for cancer that has spread to other places in the body. Central nervous systems stimulants, such as methylphenidate, may help to improve cognitive function. Physical activity uses techniques, such as aerobic and resistance exercises, which may help to improve quality of life. Giving methylphenidate and physical activity may help in reducing cancer-related fatigue in patients with metastatic cancer who receive anti-PD1 immunotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effects of methylphenidate plus physical activity (MP) compared to placebo plus physical activity (PL) in reducing cancer-related fatigue (CRF) in patients with metastatic cancer on anti-PD1 immunotherapy, as measured by changes in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) subscale scores after 2 weeks of intervention.

SECONDARY OBJECTIVES:

I. To explore the effect of MP on anxiety (Hospital Anxiety and Depression Scale [HADS]), depressed mood (HADS), cancer symptoms (Edmonton Symptom Assessment Scale (ESAS), physical activity (mean day time activity as measured by actigraphy), and serum levels of inflammatory cytokines (IL-1beta, IL-1 RA, IL-6, TNF-alpha, IL-8, IL-10, and MCP1), before and after treatment.

EXPLORATORY OBJECTIVES:

I. To determine the frequency and factors associated with CRF as assessed by FACIT-F, Patient-Reported Outcomes Measurement Information System Fatigue (PROMIS-F), Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF), actigraphy, Edmonton Symptom Assessment System (ESAS), and serum levels of inflammatory cytokines (IL-1beta, IL-1 RA, IL-6, TNF-alpha, IL-10, IL-8, MCP-1), before and during 4 initial doses of Immunotherapy.

II. To explore the effects of MP on percentage (%) of patients with dose reduction and/or discontinuation anti-PD1 immunotherapy due to CRF.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive methylphenidate orally (PO) twice daily (BID) for up to 2 weeks in the absence of disease progression or unacceptable toxicity. Patients also complete physical activity consisting of walking and resistance exercise over 25-40 minutes once daily (QD) 4 days a week. After 2 weeks, patients may continue methylphenidate at the discretion of the treating physician for up to 12 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive a matched placebo PO BID and complete physical activity as in Arm I.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: have a diagnosis of metastatic or recurrent cancer and previously received anti PD1 immunotherapy provided that they received therapy up to 1 month prior to enrollment
* Part 1: be willing to engage in follow-up telephone calls with a research staff
* Part 1: have telephone access so they can be contacted by the research staff
* Part 1: hemoglobin level of >= 8 g/dL within 2 weeks of enrollment

  * Packed red blood cell (PRBC) transfusions will be allowed to patients with hemoglobin < 8 g/dl
* Part 1: be able to understand the description of the study and give written informed consent
* Part 1: able to read, write and speak English
* Part 2: have a diagnosis of metastatic or recurrent cancer and previously received anti PD1 immunotherapy provided that they received therapy up to 1 month prior to enrollment
* Part 2: be willing to engage in follow-up telephone calls with a research staff
* Part 2: have telephone access so they can be contacted by the research staff
* Part 2: have a hemoglobin level of >=8 g/dL within 2 weeks of enrollment

  * PRBC transfusions will be allowed to patients with hemoglobin < 8 g/dl
* Part 2: be able to understand the description of the study and give written or verbal informed consent
* Part 2: able to read, write and speak English
* Part 2: presence of fatigue as defined FACIT-F subscale of =< 34 on a 0 to 52 scale (in which 52 = no fatigue and 0 = worst possible fatigue)
* Part 2: not currently taking methylphenidate, or have taken it within the previous 10 days
* Part 2: able to complete the baseline assessment forms
* Part 2: able to understand the recommendations for participation in the study
* Part 2: can be enrolled directly to part 2 independent of part 1 if on immunotherapy and having a FACIT-F fatigue =< 34, and able to complete baseline assessment and bloodwork as detailed in Part 1 at baseline and day 14 +/-3 days. Treating Oncologist should agree for participation in the intervention trial

Exclusion Criteria:

* Part 1: patients will be excluded if (1) have clinical evidence of cognitive failure as evidenced by Memorial Delirium Assessment Scale score of >= 13 at baseline completed in person, by phone, or via video-conference
* Part 2: Patients will be excluded if (1) have clinical evidence of cognitive failure as evidenced by Memorial Delirium Assessment Scale score of >= 13 at baseline completed in person, by phone, or via video-conference
* Part 2: have a major contraindication to MP (e.g., allergy/hypersensitivity to study medications or their constituents), or conditions making adherence difficult as determined by the attending physician
* Part 2: on monoamine oxidase inhibitors, tricyclic antidepressants, or clonidine
* Part 2: history of glaucoma
* Part 2: history of have severe cardiac disease (New York Heart Association functional class III or IV)
* Part 2: tachycardia and/or uncontrolled hypertension
* Part 2: currently receiving anticoagulants, anticonvulsants (phenobarbital, diphenylhydantoin, primidone), phenylbutazone, and/or tricyclic drugs (imipramine, clomipramine, or desipramine)
* Part 2: patients with Cut Down, Annoyed, Guilty and Eye Opener-Adapted to Include Drugs (CAGE-AID) >= 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the effects of methylphenidate (MP) plus physical activity in reducing cancer-related fatigue (CRF) | Up to 12 weeks
  Effects of MP to be compared to placebo plus physical activity results. To be as measured by changes in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) sub-scale scores. A t test will be used to evaluate the difference between groups unless the data appear to be non-normally distributed, in which case a Wilcoxon rank-sum test will be used to evaluate the difference between groups.

SECONDARY OUTCOMES:
Assessment of MP effects on physical activity | Up to 12 weeks
  To be measured by mean day time activity (actigraphy). To be evaluated using descriptive statistical analyses. A t test will be used to evaluate the difference between groups unless the data appear to be non-normally distributed, in which case a Wilcoxon rank-sum test will be used to evaluate the difference between groups. Will summarize percentage (%) of patients with stable CRF scores, % patients who had dose change and/ or discontinuation of anti-PD1 immunotherapy due to CRF.
Assessment of MP effects on anxiety, depressed mood, and cancer symptoms by questionnaires | Up to 5 minutes during visit
  To be assessed using statistical methods described in primary outcomes and using outcome variables including Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF) for fatigue dimensions
Assessment of MP effects on anxiety, depressed mood, and cancer symptoms by questionnaires | Up to 5 minutes during visit
  To be assessed using statistical methods described in primary outcomes and using outcome variables including Patient-Reported Outcomes Measurement Information System Fatigue (PROMIS) for fatigue dimensions
Assessment of MP effects on anxiety, depressed mood, and cancer symptoms by questionnaires | Up to 5 minutes during visit
  To be assessed using statistical methods described in primary outcomes and using outcome variables including Hospital Anxiety and Depression Scale (HADS) for anxiety/depression
Assessment of MP effects on anxiety, depressed mood, and cancer symptoms by questionnaires | Up to 5 minutes during visit
  To be assessed using statistical methods described in primary outcomes and using outcome variables including Functional Assessment of Cancer Therapy-General (FACT-G) for Quality of Life.
Assessment of MP effects on anxiety, depressed mood, and cancer symptoms by questionnaires | Up to 5 minutes during visit
  To be assessed using statistical methods described in primary outcomes and using outcome variables including Edmonton Symptom Assessment System (ESAS), (0-10 scale for sleep disturbance, fatigue, and drowsiness).

OTHER OUTCOMES:
Assessment of MP effects on levels of serum IL-1b, IL-1 RA, IL-6, TNF-a, IL-8,IL-10, and MCP1 | At weeks 2, 6, and 10
  To be assessed using blood samples obtained from participants. To be evaluated using descriptive statistical analyses. A t test will be used to evaluate the difference between groups unless the data appear to be non-normally distributed, in which case a Wilcoxon rank-sum test will be used to evaluate the difference between groups. Will summarize percentage (%) of patients with stable CRF scores, % patients who had dose change and/ or discontinuation of anti-PD1 immunotherapy due to CRF.

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org